CLINICAL TRIAL: NCT01072500
Title: The LIFE Study - Lifestyle Interventions and Independence for Elders
Acronym: LIFE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB201701066-N; 3U01AG022376-05A2S1 (NIH); U01AG022376 (NIH)
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Sedentary Lifestyle; Risk of Disability; Aging
Keywords: Aging; Physical Activity; Exercise; Sedentary Lifestyle; Mobility; Disability; Falls; Cost effectiveness; Behavioral counseling
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Activity (Active Comparator): The physical activity intervention consists primarily of walking at moderate intensity, lower extremity resistance exercises, balance exercises, stretching and behavioral counseling.
  Interventions: Behavioral: Physical Activity
- Successful Aging (Active Comparator): The successful aging intervention consists of health education seminars regarding health-related matters and upper extremity stretching exercises.
  Interventions: Behavioral: Successful Aging

INTERVENTIONS:
Behavioral: Physical Activity — The physical activity intervention consists primarily of walking at moderate intensity, lower extremity resistance exercises, balance exercises, stretching and behavioral counseling.
  Arms: Physical Activity
Behavioral: Successful Aging — The successful aging intervention consists of health education seminars regarding health-related matters and upper extremity stretching exercises.
  Other Names: Health Education
  Arms: Successful Aging

SUMMARY:
Based upon promising results from a pilot study among 424 sedentary older adults who were randomized to a physical activity intervention or a successful aging health education intervention, a Phase 3 multi-center randomized controlled trial is being conducted to compare a moderate-intensity physical activity program to a successful aging health education program in 1,600 sedentary older adults who are followed for an average of 2.7 years.

The primary aim was to assess the long-term effects of the proposed interventions on the primary outcome of major mobility disability, defined as inability to walk 400 m.

DETAILED DESCRIPTION:
As life expectancy in the United States continues to rise, the maintenance of physical independence among older Americans has emerged as a major clinical and public health priority. Efficient and reliable locomotion, or the ability to move without assistance, is a fundamental feature of human functioning. Older people who lose mobility are less likely to remain in the community, have higher rates of morbidity, mortality, and hospitalizations and experience a poorer quality of life. Several studies have shown that regular physical activity improves physical performance, but definitive evidence showing that mobility disability can be prevented was lacking. A Phase 3 randomized controlled trial was needed to fill this evidence gap.

The LIFE Study was a Phase 3, multicenter randomized controlled trial (RCT) designed to compare a moderate-intensity physical activity program to a successful aging health education program in 1,600 sedentary older persons who are followed for an average of 2.7 years. The primary outcome was major mobility disability, defined as inability to walk 400 m. Secondary outcomes include cognitive function based on the Digit Symbol Substitution Test (DSST) and the Hopkins Verbal Learning Test (HVLT); serious fall injuries; persistent mobility disability; the combined outcome of major mobility disability or death; disability in activities of daily living; and cost-effectiveness. Tertiary outcomes include the combined outcome of mild cognitive impairment or dementia, a composite measure of the cognitive assessment battery, physical performance within pre-specified subgroups defined on the basis of race, gender and baseline physical performance, sleep-wake disturbances, dyspnea, ventilatory capacity, cardiopulmonary events, and cardiovascular events.

The physical activity intervention consists primarily of walking at moderate intensity, lower extremity resistance exercises, balance exercises, stretching and behavioral counseling. The successful aging intervention consists of health education seminars regarding health-related matters and upper extremity stretching exercises. This trial provides definitive evidence regarding whether physical activity is effective and practical for preventing major mobility disability. These results will have crucial implications for public health prevention in a rapidly aging society, and will fill an important gap in knowledge for practicing evidence-based geriatric medicine. The study will also yield valuable information concerning the efficacy and effectiveness of physical activity across a broad spectrum of important health outcomes. The study will impact both clinical practice and public health policy, and will, therefore, benefit individuals and society.

The Coordinating Center was at the University of Florida and the Data Management Analysis and Quality Control Center (DMAQC) was at Wake Forest University School of Medicine. The 8 field sites participating in the LIFE Study are University of Florida, Gainesville, Florida; Northwestern University, Chicago, Illinois; Pennington Biomedical Research Center, Baton Rouge, Louisiana; University of Pittsburgh, Pittsburgh, Pennsylvania; Stanford University, Palo Alto, California; Tufts University, Boston, Massachusetts; Wake Forest University, Winston-Salem, North Carolina; and Yale University, New Haven, Connecticut.

ELIGIBILITY:
Inclusion Criteria:

1. age 70 to 89 years; (2) summary score <10 on the short physical performance battery (SPPB) (45% are <8);90 (3) sedentary lifestyle; (4) ability to complete the 400 m walk test without an assistive device; and (5) willingness to be randomized to either intervention group.

   Exclusion Criteria:

   Exclusion Criteria for Factors that May Limit Adherence to Interventions or Affect Conduct of the Trial • Unable or unwilling to give informed consent or accept randomization in either study group • Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
   * Current consumption of more than 14 alcoholic drinks per week
   * Plans to relocate to out of the study area within the next 2 years or plans to be out of the study area for more than 6 consecutive weeks in the next year
   * Self-reported inability to walk across a small room
   * The use of a walker to complete the 400 m walk and/or unable to complete the 400 m walk without sitting down or the help of another person
   * Another member of the household is a participant in the Life Study
   * Residence too far from the intervention site
   * Residence in a nursing home
   * Difficulty in communication with study personnel due to speech or hearing problems
   * Modified Mini-Mental State Exam (3MSE) score below the cutoff for education:

   African American, 9+ yrs 76, <9 yrs 70; English Speaking Non-African American, 9+ yrs 80, <9 yrs 76; Spanish Speaking, 9+ yrs 80, <9 yrs 70
   * Participation in LIFE-Pilot study
   * Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

   Exclusion Criteria for Underlying Diseases Likely to Limit Lifespan and/or Affect the Safety of the Interventions

   • Severe arthritis (either osteoarthritis or rheumatoid arthritis)

   • Cancer requiring treatment in the past three years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer)

   • Lung disease requiring either regular use of corticosteroid pills or injections or the use of supplemental oxygen

   • Development of chest pain or severe shortness of breath on a 400 m self-paced walk test

   • Cardiovascular disease (including New York Heart Association Class III or IV congestive heart failure, clinically significant aortic stenosis, history or cardiac arrest, use of a cardiac defibrillator or uncontrolled angina)

   • Parkinson's disease or other serious neurological disorder

   • Renal disease requiring dialysis

   • Other illness of such severity that life expectancy is considered to be less than 12 months

   • Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the clinical site

   Temporary Exclusion Criteria

   • Uncontrolled hypertension (systolic blood pressure > 200 mmHg and/or diastolic blood pressure > 110 mmHg).

   • Uncontrolled diabetes with recent weight loss, diabetic coma or frequent insulin reactions.
   * Stroke, hip fracture, hip or knee replacement, or spinal surgery in the past 6 months.
   * Serious conduction disorder (e.g., 3rd degree heart block), uncontrolled arrhythmia, or new Q waves or ST-segment depressions (>3 mm) on ECG.
   * Myocardial infarction, major heart surgery (i.e., valve replacement or bypass surgery), stroke, deep vein thrombosis or pulmonary embolus in the past 6 months.
   * Undergoing physical therapy or cardiopulmonary rehabilitation
   * Currently enrolled in another randomized trial involving lifestyle or pharmaceutical interventions

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1635 (Actual)
Dates: Start 2010-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pahor, MD, Principal Investigator — University of Florida
Locations (8):
- United States (8):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Pennington Biodmedical Research, Baton Rouge, Louisiana
  - Tufts University, Boston, Massachusetts
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
If an investigator outside of a LIFE study team would like access to the LIFE coded dataset, this individual must go through the following steps:
  1. Request access to the LIFE website for the purposes of submitting a P&P proposal to obtain access to the Coded Datasets by going to the LIFE website (www.thelifestudy.org) and clicking on the button "Request for Non-LIFE investigator Access" and completing the request form.
  2. Access would be granted to the LIFE website where access to would be provided to the data dictionary, data documentation, and protocol, in addition to the Manuscript Proposal Submission Form.
  3. A proposal would be submitted (per current guidelines) to LIFE and reviewed through the usual channels.
  4. If approved the Investigator would be sent a Coded Data Use Agreement document to be signed and sent back to the DMAQC for filing.
  5. Access to the Coded Datasets would be granted for a period of 10 days.

REFERENCES:
- [Background] LIFE Study Investigators; Pahor M, Blair SN, Espeland M, Fielding R, Gill TM, Guralnik JM, Hadley EC, King AC, Kritchevsky SB, Maraldi C, Miller ME, Newman AB, Rejeski WJ, Romashkan S, Studenski S. Effects of a physical activity intervention on measures of physical performance: Results of the lifestyle interventions and independence for Elders Pilot (LIFE-P) study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1157-65. doi: 10.1093/gerona/61.11.1157. PMID 17167156
- [Background] Fielding RA, Rejeski WJ, Blair S, Church T, Espeland MA, Gill TM, Guralnik JM, Hsu FC, Katula J, King AC, Kritchevsky SB, McDermott MM, Miller ME, Nayfield S, Newman AB, Williamson JD, Bonds D, Romashkan S, Hadley E, Pahor M; LIFE Research Group. The Lifestyle Interventions and Independence for Elders Study: design and methods. J Gerontol A Biol Sci Med Sci. 2011 Nov;66(11):1226-37. doi: 10.1093/gerona/glr123. Epub 2011 Aug 8. PMID 21825283
- [Result] Rejeski WJ, Marsh AP, Anton S, Chen SH, Church T, Gill TM, Guralnik JM, Glynn NW, King AC, Rushing J, Ip EH; LIFE Research Group. The MAT-sf: clinical relevance and validity. J Gerontol A Biol Sci Med Sci. 2013 Dec;68(12):1567-74. doi: 10.1093/gerona/glt068. Epub 2013 May 17. PMID 23685766
- [Result] Espeland MA, Katula JA, Rushing J, Kramer AF, Jennings JM, Sink KM, Nadkarni NK, Reid KF, Castro CM, Church T, Kerwin DR, Williamson JD, Marottoli RA, Rushing S, Marsiske M, Rapp SR; LIFE Study Group. Performance of a computer-based assessment of cognitive function measures in two cohorts of seniors. Int J Geriatr Psychiatry. 2013 Dec;28(12):1239-50. doi: 10.1002/gps.3949. Epub 2013 Apr 16. PMID 23589390
- [Result] Marsh AP, Lovato LC, Glynn NW, Kennedy K, Castro C, Domanchuk K, McDavitt E, Rodate R, Marsiske M, McGloin J, Groessl EJ, Pahor M, Guralnik JM; LIFE Study Research Group. Lifestyle interventions and independence for elders study: recruitment and baseline characteristics. J Gerontol A Biol Sci Med Sci. 2013 Dec;68(12):1549-58. doi: 10.1093/gerona/glt064. Epub 2013 May 28. PMID 23716501
- [Result] McDermott MM, Applegate WB, Bonds DE, Buford TW, Church T, Espeland MA, Gill TM, Guralnik JM, Haskell W, Lovato LC, Pahor M, Pepine CJ, Reid KF, Newman A. Ankle brachial index values, leg symptoms, and functional performance among community-dwelling older men and women in the lifestyle interventions and independence for elders study. J Am Heart Assoc. 2013 Nov 12;2(6):e000257. doi: 10.1161/JAHA.113.000257. PMID 24222666
- [Result] Rejeski WJ, Axtell R, Fielding R, Katula J, King AC, Manini TM, Marsh AP, Pahor M, Rego A, Tudor-Locke C, Newman M, Walkup MP, Miller ME; LIFE Study Investigator Group. Promoting physical activity for elders with compromised function: the lifestyle interventions and independence for elders (LIFE) study physical activity intervention. Clin Interv Aging. 2013;8:1119-31. doi: 10.2147/CIA.S49737. Epub 2013 Sep 12. PMID 24049442
- [Derived] Levati E, Zazzara MB, Iurlaro A, Marzetti E, Calvani R, Pahor M, Picca A, Tosato M, Landi F, Bernabei R, Onder G. Lifestyle interventions and medication burden in older adults: insights from the Lifestyle Intervention and Independence for Elders (LIFE) and the Sarcopenia and Physical fRailty iN older people: multi-componenT Treatment strategies (SPRINTT) trials. Eur Geriatr Med. 2025 Oct;16(5):1591-1598. doi: 10.1007/s41999-025-01266-0. Epub 2025 Jul 15. PMID 40665144
- [Derived] Fielding RA, Atkinson EJ, Aversa Z, White TA, Heeren AA, Mielke MM, Cummings SR, Pahor M, Leeuwenburgh C, LeBrasseur NK. Biomarkers of Cellular Senescence Predict the Onset of Mobility Disability and Are Reduced by Physical Activity in Older Adults. J Gerontol A Biol Sci Med Sci. 2024 Mar 1;79(3):glad257. doi: 10.1093/gerona/glad257. PMID 37948612
- [Derived] Custodero C, Agosti P, Anton SD, Manini TM, Lozupone M, Panza F, Pahor M, Sabba C, Solfrizzi V. Effect of Physical Activity Intervention on Gait Speed by Frailty Condition: A Randomized Clinical Trial. J Am Med Dir Assoc. 2023 Apr;24(4):489-496. doi: 10.1016/j.jamda.2023.01.023. Epub 2023 Mar 3. PMID 36878264
- [Derived] Fielding RA, Atkinson EJ, Aversa Z, White TA, Heeren AA, Achenbach SJ, Mielke MM, Cummings SR, Pahor M, Leeuwenburgh C, LeBrasseur NK. Associations between biomarkers of cellular senescence and physical function in humans: observations from the lifestyle interventions for elders (LIFE) study. Geroscience. 2022 Dec;44(6):2757-2770. doi: 10.1007/s11357-022-00685-2. Epub 2022 Nov 11. PMID 36367600
- [Derived] Shlipak MG, Sheshadri A, Hsu FC, Chen SH, Jotwani V, Tranah G, Fielding RA, Liu CK, Ix J, Coca SG; LIFE Investigators. Effect of Structured, Moderate Exercise on Kidney Function Decline in Sedentary Older Adults: An Ancillary Analysis of the LIFE Study Randomized Clinical Trial. JAMA Intern Med. 2022 Jun 1;182(6):650-659. doi: 10.1001/jamainternmed.2022.1449. PMID 35499834
- [Derived] Botoseneanu A, Chen H, Ambrosius WT, Allore HG, Anton S, Folta SC, King AC, Nicklas BJ, Spring B, Strotmeyer ES, Gill TM. Metabolic syndrome and the benefit of a physical activity intervention on lower-extremity function: Results from a randomized clinical trial. Exp Gerontol. 2021 Jul 15;150:111343. doi: 10.1016/j.exger.2021.111343. Epub 2021 Apr 10. PMID 33848565
- [Derived] Fanning J, Rejeski WJ, Chen SH, Guralnik J, Pahor M, Miller ME. Relationships Between Profiles of Physical Activity and Major Mobility Disability in the LIFE Study. J Am Geriatr Soc. 2020 Jul;68(7):1476-1483. doi: 10.1111/jgs.16386. Epub 2020 Mar 20. PMID 32196636
- [Derived] Fanning J, Rejeski WJ, Chen SH, Nicklas BJ, Walkup MP, Axtell RS, Fielding RA, Glynn NW, King AC, Manini TM, McDermott MM, Newman AB, Pahor M, Tudor-Locke C, Miller ME; LIFE Study Investigators. A Case for Promoting Movement Medicine: Preventing Disability in the LIFE Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2019 Oct 4;74(11):1821-1827. doi: 10.1093/gerona/glz050. PMID 30778518
- [Derived] Liu Z, Hsu FC, Trombetti A, King AC, Liu CK, Manini TM, Fielding RA, Pahor M, Newman AB, Kritchevsky S, Gill TM; LIFE Study investigators. Effect of 24-month physical activity on cognitive frailty and the role of inflammation: the LIFE randomized clinical trial. BMC Med. 2018 Oct 24;16(1):185. doi: 10.1186/s12916-018-1174-8. PMID 30352583
- [Derived] Datta R, Trentalange M, Van Ness PH, McGloin JM, Guralnik JM, Miller ME, Walkup MP, Nadkarni N, Pahor M, Gill TM, Quagliarello V, Juthani-Mehta M; LIFE Study Group. Serious adverse events of older adults in nursing home and community intervention trials. Contemp Clin Trials Commun. 2017 Dec 21;9:77-80. doi: 10.1016/j.conctc.2017.12.004. eCollection 2018 Mar. PMID 29696228
- [Derived] Rosso AL, Metti AL, Glynn NW, Boudreau RM, Rejeski WJ, Bohnen N, Chen H, Johannsen NM, King AC, Manini TM, Pahor M, Studenski SA, Fragoso CAV, Rosano C; LIFE Study Group. Dopamine-Related Genotypes and Physical Activity Change During an Intervention: The Lifestyle Interventions and Independence for Elders Study. J Am Geriatr Soc. 2018 Jul;66(6):1172-1179. doi: 10.1111/jgs.15369. Epub 2018 Apr 10. PMID 29637543
- [Derived] Cochrane SK, Chen SH, Fitzgerald JD, Dodson JA, Fielding RA, King AC, McDermott MM, Manini TM, Marsh AP, Newman AB, Pahor M, Tudor-Locke C, Ambrosius WT, Buford TW; LIFE Study Research Group. Association of Accelerometry-Measured Physical Activity and Cardiovascular Events in Mobility-Limited Older Adults: The LIFE (Lifestyle Interventions and Independence for Elders) Study. J Am Heart Assoc. 2017 Dec 2;6(12):e007215. doi: 10.1161/JAHA.117.007215. PMID 29197830
- [Derived] Kritchevsky SB, Lovato L, Handing EP, Blair S, Botoseneanu A, Guralnik JM, Liu C, King A, Marsh AP, Pahor M, Rejeski WJ, Spring B, Manini T. Exercise's effect on mobility disability in older adults with and without obesity: The LIFE study randomized clinical trial. Obesity (Silver Spring). 2017 Jul;25(7):1199-1205. doi: 10.1002/oby.21860. PMID 28653499
- [Derived] Gill TM, Beavers DP, Guralnik JM, Pahor M, Fielding RA, Hauser M, Manini TM, Marsh AP, McDermott MM, Newman AB, Allore HG, Miller ME; LIFE Study Investigators. The effect of intervening hospitalizations on the benefit of structured physical activity in promoting independent mobility among community-living older persons: secondary analysis of a randomized controlled trial. BMC Med. 2017 Mar 28;15(1):65. doi: 10.1186/s12916-017-0824-6. PMID 28347337
- [Derived] King AC, Salvo D, Banda JA, Ahn DK, Chapman JE, Gill TM, Fielding RA, Demons J, Tudor-Locke C, Rosso A, Pahor M, Frank LD. Preserving older adults' routine outdoor activities in contrasting neighborhood environments through a physical activity intervention. Prev Med. 2017 Mar;96:87-93. doi: 10.1016/j.ypmed.2016.12.049. Epub 2016 Dec 28. PMID 28039068
- [Derived] O Hartaigh B, Lovato LC, Pahor M, Buford TW, Dodson JA, Forman DE, Buman MP, Demons JL, Santanasto AJ, Liu C, Miller ME, McDermott MM, Gill TM; LIFE Study Group. Effect of a Long-Term Physical Activity Intervention on Resting Pulse Rate in Older Persons: Results from the Lifestyle Interventions and Independence for Elders Study. J Am Geriatr Soc. 2016 Dec;64(12):2511-2516. doi: 10.1111/jgs.14380. Epub 2016 Oct 27. PMID 27787876
- [Derived] Gill TM, Guralnik JM, Pahor M, Church T, Fielding RA, King AC, Marsh AP, Newman AB, Pellegrini CA, Chen SH, Allore HG, Miller ME; LIFE Study Investigators. Effect of Structured Physical Activity on Overall Burden and Transitions Between States of Major Mobility Disability in Older Persons: Secondary Analysis of a Randomized Trial. Ann Intern Med. 2016 Dec 20;165(12):833-840. doi: 10.7326/M16-0529. Epub 2016 Sep 27. PMID 27669457
- [Derived] Marsh AP, Applegate WB, Guralnik JM, Jack Rejeski W, Church TS, Fielding RA, Gill TM, King AC, Kritchevsky SB, Manini TM, McDermott MM, Newman AB, Stowe CL, Walkup MP, Pahor M, Miller ME; LIFE Study Investigators. Hospitalizations During a Physical Activity Intervention in Older Adults at Risk of Mobility Disability: Analyses from the Lifestyle Interventions and Independence for Elders Randomized Clinical Trial. J Am Geriatr Soc. 2016 May;64(5):933-43. doi: 10.1111/jgs.14114. PMID 27225353
- [Derived] Bann D, Chen H, Bonell C, Glynn NW, Fielding RA, Manini T, King AC, Pahor M, Mihalko SL, Gill TM; Life Study investigators. Socioeconomic differences in the benefits of structured physical activity compared with health education on the prevention of major mobility disability in older adults: the LIFE study. J Epidemiol Community Health. 2016 Sep;70(9):930-3. doi: 10.1136/jech-2016-207321. Epub 2016 Apr 8. PMID 27060177
- [Derived] Vaz Fragoso CA, Beavers DP, Anton SD, Liu CK, McDermott MM, Newman AB, Pahor M, Stafford RS, Gill TM; Lifestyle Interventions and Independence in Elders Investigators. Effect of Structured Physical Activity on Respiratory Outcomes in Sedentary Elderly Adults with Mobility Limitations. J Am Geriatr Soc. 2016 Mar;64(3):501-9. doi: 10.1111/jgs.14013. PMID 27000324
- [Derived] Groessl EJ, Kaplan RM, Castro Sweet CM, Church T, Espeland MA, Gill TM, Glynn NW, King AC, Kritchevsky S, Manini T, McDermott MM, Reid KF, Rushing J, Pahor M; LIFE Study Group. Cost-effectiveness of the LIFE Physical Activity Intervention for Older Adults at Increased Risk for Mobility Disability. J Gerontol A Biol Sci Med Sci. 2016 May;71(5):656-62. doi: 10.1093/gerona/glw001. Epub 2016 Feb 17. PMID 26888433
- [Derived] Gill TM, Pahor M, Guralnik JM, McDermott MM, King AC, Buford TW, Strotmeyer ES, Nelson ME, Sink KM, Demons JL, Kashaf SS, Walkup MP, Miller ME; LIFE Study Investigators. Effect of structured physical activity on prevention of serious fall injuries in adults aged 70-89: randomized clinical trial (LIFE Study). BMJ. 2016 Feb 3;352:i245. doi: 10.1136/bmj.i245. PMID 26842425
- [Derived] King AC, Salvo D, Banda JA, Ahn DK, Gill TM, Miller M, Newman AB, Fielding RA, Siordia C, Moore S, Folta S, Spring B, Manini T, Pahor M; LIFE Study Investigators. An observational study identifying obese subgroups among older adults at increased risk of mobility disability: do perceptions of the neighborhood environment matter? Int J Behav Nutr Phys Act. 2015 Dec 18;12:157. doi: 10.1186/s12966-015-0322-1. PMID 26684894
- [Derived] Sink KM, Espeland MA, Castro CM, Church T, Cohen R, Dodson JA, Guralnik J, Hendrie HC, Jennings J, Katula J, Lopez OL, McDermott MM, Pahor M, Reid KF, Rushing J, Verghese J, Rapp S, Williamson JD; LIFE Study Investigators. Effect of a 24-Month Physical Activity Intervention vs Health Education on Cognitive Outcomes in Sedentary Older Adults: The LIFE Randomized Trial. JAMA. 2015 Aug 25;314(8):781-90. doi: 10.1001/jama.2015.9617. PMID 26305648
- [Derived] Vaz Fragoso CA, Miller ME, King AC, Kritchevsky SB, Liu CK, Myers VH, Nadkarni NK, Pahor M, Spring BJ, Gill TM; Lifestyle Interventions and Independence for Elders Study Group. Effect of Structured Physical Activity on Sleep-Wake Behaviors in Sedentary Elderly Adults with Mobility Limitations. J Am Geriatr Soc. 2015 Jul;63(7):1381-90. doi: 10.1111/jgs.13509. Epub 2015 Jun 26. PMID 26115386
- [Derived] Espeland MA, Newman AB, Sink K, Gill TM, King AC, Miller ME, Guralnik J, Katula J, Church T, Manini T, Reid KF, McDermott MM; LIFE Study Group. Associations Between Ankle-Brachial Index and Cognitive Function: Results From the Lifestyle Interventions and Independence for Elders Trial. J Am Med Dir Assoc. 2015 Aug 1;16(8):682-9. doi: 10.1016/j.jamda.2015.03.010. Epub 2015 Apr 11. PMID 25869993
- [Derived] Fitzgerald JD, Johnson L, Hire DG, Ambrosius WT, Anton SD, Dodson JA, Marsh AP, McDermott MM, Nocera JR, Tudor-Locke C, White DK, Yank V, Pahor M, Manini TM, Buford TW; LIFE Study Research Group. Association of objectively measured physical activity with cardiovascular risk in mobility-limited older adults. J Am Heart Assoc. 2015 Feb 18;4(2):e001288. doi: 10.1161/JAHA.114.001288. PMID 25696062
- [Derived] Bann D, Hire D, Manini T, Cooper R, Botoseneanu A, McDermott MM, Pahor M, Glynn NW, Fielding R, King AC, Church T, Ambrosius WT, Gill TM; LIFE Study Group. Light Intensity physical activity and sedentary behavior in relation to body mass index and grip strength in older adults: cross-sectional findings from the Lifestyle Interventions and Independence for Elders (LIFE) study. PLoS One. 2015 Feb 3;10(2):e0116058. doi: 10.1371/journal.pone.0116058. eCollection 2015. PMID 25647685
- [Derived] Vaz Fragoso CA, Hsu FC, Brinkley T, Church T, Liu CK, Manini T, Newman AB, Stafford RS, McDermott MM, Gill TM; LIFE Study Group. Combined reduced forced expiratory volume in 1 second (FEV1) and peripheral artery disease in sedentary elders with functional limitations. J Am Med Dir Assoc. 2014 Sep;15(9):665-70. doi: 10.1016/j.jamda.2014.05.008. Epub 2014 Jun 25. PMID 24973990
- [Derived] Vaz Fragoso CA, Miller ME, Fielding RA, King AC, Kritchevsky SB, McDermott MM, Myers V, Newman AB, Pahor M, Gill TM; Lifestyle Interventions and Independence in Elder Study Group. Sleep-wake disturbances in sedentary community-dwelling elderly adults with functional limitations. J Am Geriatr Soc. 2014 Jun;62(6):1064-72. doi: 10.1111/jgs.12845. Epub 2014 Jun 2. PMID 24889836
- [Derived] Pahor M, Guralnik JM, Ambrosius WT, Blair S, Bonds DE, Church TS, Espeland MA, Fielding RA, Gill TM, Groessl EJ, King AC, Kritchevsky SB, Manini TM, McDermott MM, Miller ME, Newman AB, Rejeski WJ, Sink KM, Williamson JD; LIFE study investigators. Effect of structured physical activity on prevention of major mobility disability in older adults: the LIFE study randomized clinical trial. JAMA. 2014 Jun 18;311(23):2387-96. doi: 10.1001/jama.2014.5616. PMID 24866862
- [Derived] Vaz Fragoso CA, Beavers DP, Hankinson JL, Flynn G, Berra K, Kritchevsky SB, Liu CK, McDermott MM, Manini TM, Rejeski WJ, Gill TM; Lifestyle Interventions Independence for Elders Study Investigators. Respiratory impairment and dyspnea and their associations with physical inactivity and mobility in sedentary community-dwelling older persons. J Am Geriatr Soc. 2014 Apr;62(4):622-8. doi: 10.1111/jgs.12738. Epub 2014 Mar 17. PMID 24635756
- See also: The LIFE Study website — http://www.thelifestudy.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1,635 participants were randomized over 21-months, with the target of 1,600 reached late Nov 2011. The 1st randomization occurred 3/12/10, and the final randomization on 12/27/11. Participants in the recruitment pipeline completed screening and testing visits and were randomized; hence, the total randomized exceeded the target.
Groups:
- Successful Aging (Health Education): The successful aging intervention consists of health education seminars regarding health-related matters and upper extremity stretching exercises.
Period: Overall Study
Arm/Group | Physical Activity | Successful Aging (Health Education)
Started | 818 | 817
Completed | 794 | 803
Not Completed | 24 | 14
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 17 | 10

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were similar in the 2 groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity | Successful Aging | Total
Number analyzed (Participants) | 818 | 817 | 1635
Age, Continuous [Mean (Standard Deviation); unit: years] — These represent data that was measured and analyzed. We have verified the standard deviation is the same in both arms.
  years | 78.7 (5.2) | 79.1 (5.2) | 78.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 547 | 551 | 1098
  Male | 271 | 266 | 537
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 31 | 30 | 61
  White | 604 | 635 | 1239
  African American | 163 | 125 | 288
  Asian | 7 | 8 | 15
  Other/Mixed | 10 | 17 | 27
  Refused/Missing | 3 | 2 | 5
Education [Number; unit: participants]
  No formal eduction | 7 | 6 | 13
  Elementary School (k-8) | 15 | 17 | 32
  High school/equivalent (9-12) | 248 | 236 | 484
  College (13-17) | 321 | 320 | 641
  Post Graduate | 194 | 208 | 402
  Other | 32 | 26 | 58
  Unknown | 1 | 4 | 5
Total SPPB Score [Mean (Standard Deviation); unit: units on a scale] — This is the Short Physical Performance Battery with a Scale from 0-12. Lower scores represent worse physical performance. Three subscales (balance, gait speed, and chair stand) are summed to create the total score.
  units on a scale | 7.4 (1.6) | 7.3 (1.6) | 7.4 (1.6)
3MSE Score, 0-100 scale, mean [Mean (Standard Deviation); unit: units on a scale] — Modified Mini-Mental State Exam Higher scores indicate better cognition score
  units on a scale | 91.5 (5.6) | 91.6 (5.5) | 91.5 (5.5)
CHAMPS 18 Total Score [Mean (Standard Deviation); unit: hours/week] — Community Health Activities Model Program for Seniors - Activity Questionnaire Score is based on hours of moderate-intensity exercise-related activities per week (frequency/week) Total score is the sum of each activity's frequency. The minimum total score is 0 and the maximum is 168.
  hours/week | 15.9 (32.1) | 18.2 (33.8) | 17.0 (33.0)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 179.3 (39.6) | 178.5 (39.9) | 178.9 (39.8)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — mean of two measures
  mmHg | 127.9 (18.1) | 127.0 (17.8) | 127.4 (18.0)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — mean of two measures
  mmHg | 68.7 (10.3) | 67.7 (10.1) | 68.2 (10.2)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 81.9 (18.4) | 82.0 (19.3) | 81.9 (18.8)
Body Mass Index, mean [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (5.9) | 30.3 (6.2) | 30.2 (6.1)
High blood pressure/hypertension [Number; unit: participants] — The number of participants in this measurement (high blood pressure) are the ones who self-reported this history.
  participants | 573 | 578 | 1151
Heart Attack/Coronary/MI [Number; unit: participants] — The number of participants in this measurement (heart attack/coronary/MI) are the ones who self-reported this history.
  participants | 60 | 69 | 129
Heart failure/congestive heart failure [Number; unit: participants] — The number of participants in this measurement (heart failure/congestive heart failure) are the ones who self-reported this history.
  participants | 26 | 45 | 71
Pacemaker [Number; unit: participants] — The number of participants in this measurement (pacemaker) are the ones who self-reported this history.
  participants | 33 | 33 | 66
Stroke [Number; unit: participants] — The number of participants in this measurement (stroke) are the ones who self-reported this history.
  participants | 57 | 52 | 109
Cancer [Number; unit: participants] — The number of participants in this measurement (cancer) are the ones who self-reported this history.
  participants | 178 | 192 | 370
Diabetes/High Blood Sugar [Number; unit: participants] — The number of participants in this measurement (diabetes/high blood sugar) are the ones who self-reported this history.
  participants | 198 | 216 | 414
Chronic lung disease [Number; unit: participants] — The number of participants in this measurement (chronic lung disease) are the ones who self-reported this history.
  participants | 130 | 123 | 253

OUTCOME MEASURES:

1. Primary Outcome: Major Mobility Disability, Defined as Incapacity to Walk 400 Meters
Description: The primary outcome of major mobility disability was defined as the inability to complete a 400-m walk test within 15 minutes without sitting and without the help of another person or walker. Use of a cane was acceptable. Participants were asked to walk 400 m at their usual pace, without overexerting, on a 20 meter course for 10 laps (40 meters/lap). Participants were allowed to stop for up to 1 minute for fatigue or related symptoms. When major mobility disability could not be objectively measured because of the inability of the participant to come to the clinic and absence of a suitable walking course at the participant's home, institution, or hospital, an alternative adjudication of the outcome was based on objective inability to walk 4 meters in less than 10 seconds, or self-, proxy-, or medical record-reported inability to walk across a room. If participants met these alternative criteria, they would not be able to complete the 400 meter walk within 15 minutes.
Time Frame: Median 2.7 years/Average 2.6 years
Measure: Number; unit: participants
Arm/Group | Physical Activity | Successful Aging
Number analyzed (Participants) | 818 | 817
participants | 246 | 290
Statistical Analysis 1: Comparison: Physical Activity vs Successful Aging; Test type: Superiority or Other; p = 0.03, Regression, Cox; To compare interventions, we used a likelihood ratio test from a Cox regression model, stratified by field center and sex; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.69 to 0.98]

2. Secondary Outcome: Persistent Mobility Disability (Assessed Every 6 Months)
Description: The assessment of major mobility disability (the inability to complete a 400-m walk test within 15 minutes without sitting and without the help of another person or walker. Use of a cane was acceptable. Participants were asked to walk 400m at their usual pace, without overexerting, on a 20 meter course for 10 laps (40 meters/lap). Participants were allowed to stop for up to 1 minute for fatigue or related symptoms. When MMD could not be objectively measured because of the inability of the participant to come to the clinic and absence of a suitable walking course at the participant's home, institution, or hospital, an alternative adjudication of the outcome was based on objective inability to walk 4 meters in less than 10 seconds, or self-, proxy-, or medical record-reported inability to walk across a room. If participants met these alternative criteria, they would not be able to complete the 400 m walk within 15 minutes.) at two consecutive time points or MMD followed by death.
Time Frame: Median 2.7 years/Average 2.6 years
Measure: Number; unit: participants
Arm/Group | Physical Activity | Successful Aging
Number analyzed (Participants) | 818 | 817
participants | 120 | 162
Statistical Analysis 1: Comparison: Physical Activity vs Successful Aging; Test type: Superiority or Other; p = 0.006, Regression, Cox; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.57 to 0.91]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from each participant beginning with screening until closeout of the study. Participants were queried every 6 months but could report adverse events in-between visits. Participants were followed for an average of 2.6 years.
Description: To minimize reporting bias, adverse events originating from the blinded assessments are presented. Blinded assessments were completed every 6 months.
  Non-serious AEs were collected without regard to the specific AE term.
Arm/Group | Physical Activity | Successful Aging
Serious Adverse Events (participants affected / at risk) | 404/818 | 373/817
Other Adverse Events (participants affected / at risk) | 181/818 | 88/817
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity (N=818) | Successful Aging (N=817)
ABDOMINAL INFECTION (Infections and infestations) | 0 (0) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 (12) | 6 (7)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 6 (6) | 6 (6)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 4 (5) | 4 (4)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (2) | 0 (0)
ALLERGIC REACTION (Immune system disorders) | 5 (7) | 1 (1)
ANAPHYLAXIS (Immune system disorders) | 0 (0) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 10 (15) | 6 (6)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
ANORECTAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
AORTIC VALVE DISEASE (Cardiac disorders) | 3 (3) | 2 (2)
APNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 1 (1)
APPENDICITIS PERFORATED (Infections and infestations) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 14 (15) | 15 (15)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
ASYSTOLE (Cardiac disorders) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 2 (3) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 23 (28) | 19 (23)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 2 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (7)
BILIARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BLADDER INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
BONE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
BRONCHIAL INFECTION (Infections and infestations) | 8 (9) | 4 (4)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 6 (6) | 7 (7)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 11 (11) | 8 (8)
CATHETER RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CENTRAL NERVOUS SYSTEM NECROSIS (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROSPINAL FLUID LEAKAGE (Nervous system disorders) | 0 (0) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 18 (24) | 12 (14)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
CHOLECYSTITIS (Hepatobiliary disorders) | 3 (3) | 2 (2)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1) | 0 (0)
COGNITIVE DISTURBANCE (Nervous system disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 4 (4) | 3 (3)
COLONIC FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLONIC HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 0 (0)
COLONIC PERFORATION (Gastrointestinal disorders) | 1 (1) | 2 (2)
CONDUCTION DISORDER (Cardiac disorders) | 1 (1) | 2 (2)
CONFUSION (Psychiatric disorders) | 0 (0) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 1 (2) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
DEATH NOS (General disorders) | 4 (4) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 12 (12) | 9 (9)
DELIRIUM (Psychiatric disorders) | 2 (2) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 3 (3) | 4 (4)
DIZZINESS (Nervous system disorders) | 10 (11) | 5 (5)
DYSESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 3 (3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 7 (8)
EDEMA LIMBS (General disorders) | 0 (0) | 3 (3)
EDEMA TRUNK (General disorders) | 0 (0) | 1 (1)
ENCEPHALITIS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 1 (1) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0)
ESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
FACIAL MUSCLE WEAKNESS (Nervous system disorders) | 1 (1) | 0 (0)
FACIAL NERVE DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 28 (29) | 31 (35)
FATIGUE (General disorders) | 3 (3) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (4)
FEVER (General disorders) | 1 (5) | 1 (2)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 3 (3)
FRACTURE (Injury, poisoning and procedural complications) | 18 (19) | 19 (19)
GAIT DISTURBANCE (General disorders) | 1 (2) | 0 (0)
GALLBLADDER INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GALLBLADDER NECROSIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
GALLBLADDER OBSTRUCTION (Hepatobiliary disorders) | 2 (2) | 1 (1)
GALLBLADDER PAIN (Hepatobiliary disorders) | 2 (2) | 1 (1)
GASTRIC HEMORRHAGE (Gastrointestinal disorders) | 4 (4) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 2 (2) | 4 (5)
GASTRITIS (Gastrointestinal disorders) | 2 (2) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 5 (8) | 3 (3)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 31 (49) | 27 (46)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
HALLUCINATIONS (Psychiatric disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
HEART FAILURE (Cardiac disorders) | 20 (24) | 16 (23)
HEMATOMA (Vascular disorders) | 3 (3) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 1 (1) | 3 (3)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (2) | 0 (0)
HEPATIC HEMORRHAGE (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 1 (1) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
HYDROCEPHALUS (Nervous system disorders) | 1 (1) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
HYPERKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPERPARATHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 6 (7) | 8 (8)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOPARATHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 8 (8) | 5 (5)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ILEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (1)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 0 (0) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 6 (6) | 1 (1)
INJECTION SITE REACTION (General disorders) | 1 (1) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INR INCREASED (Investigations) | 0 (0) | 1 (1)
INTRA-ABDOMINAL HEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 0 (0)
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 4 (5) | 3 (4)
INTRAOPERATIVE CARDIAC INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ISCHEMIA CEREBROVASCULAR (Nervous system disorders) | 0 (0) | 2 (3)
JEJUNAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
JOINT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
JOINT RANGE OF MOTION DECREASED CERVICAL SPINE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
JOINT RANGE OF MOTION DECREASED LUMBAR SPINE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 1 (1) | 1 (1)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1)
LOWER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 2 (3) | 1 (1)
LUNG INFECTION (Infections and infestations) | 15 (17) | 15 (16)
MALAISE (General disorders) | 0 (0) | 1 (1)
MANIA (Psychiatric disorders) | 1 (1) | 0 (0)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 9 (9) | 17 (18)
MUSCULOSKELETAL DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 14 (14) | 12 (13)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 (31) | 19 (31)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 4 (5) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 11 (11) | 8 (9)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
OVARIAN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (9)
PALPITATIONS (Cardiac disorders) | 1 (2) | 1 (1)
PANCREATIC NECROSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 2 (2) | 5 (5)
PAROXYSMAL ATRIAL TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDITIS (Cardiac disorders) | 1 (1) | 1 (1)
PERIPHERAL ISCHEMIA (Vascular disorders) | 2 (3) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 2 (3) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 17 (23) | 11 (11)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 5 (6) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PROSTATE INFECTION (Infections and infestations) | 1 (1) | 1 (1)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 2 (2) | 0 (0)
PROSTECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
RADICULITIS (Nervous system disorders) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 2 (3)
RECTAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 1 (1) | 5 (5)
RENAL CALCULI (Renal and urinary disorders) | 3 (3) | 2 (2)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY (Reproductive system and breast disorders) | 1 (1) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 4 (5)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (9)
RESTRICTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
SALIVARY GLAND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 3 (4) | 2 (2)
SEPSIS (Infections and infestations) | 7 (7) | 3 (3)
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 3 (3) | 7 (7)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5)
SKIN INFECTION (Infections and infestations) | 6 (6) | 7 (9)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 8 (8) | 2 (2)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SOFT TISSUE NECROSIS UPPER LIMB (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
STOMACH PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2)
STROKE (Nervous system disorders) | 15 (19) | 22 (25)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 67 (75) | 74 (86)
SYNCOPE (Nervous system disorders) | 13 (15) | 15 (17)
THROMBOEMBOLIC EVENT (Vascular disorders) | 11 (12) | 10 (12)
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 10 (10) | 8 (9)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
TUMOR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 2 (2) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 2 (2) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 11 (11) | 13 (14)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT PAIN (Renal and urinary disorders) | 0 (0) | 2 (2)
UTERINE PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL HEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 5 (6) | 3 (3)
VASOVAGAL REACTION (Nervous system disorders) | 1 (1) | 0 (0)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 (3) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 5 (5) | 6 (6)
VISCERAL ARTERIAL ISCHEMIA (Vascular disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 4 (6) | 3 (3)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
WHITE BLOOD CELL DECREASED (Investigations) | 0 (0) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 2 (2) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity (N=818) | Successful Aging (N=817)
non-serious AES (General disorders) | 181 (181) | 88 (88)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No